CLINICAL TRIAL: NCT05747755
Title: Achieving Diagnostic Excellence Through Prevention and Teamwork (ADEPT)
Brief Title: Achieving Diagnostic Excellence Through Prevention and Teamwork
Acronym: ADEPT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Jeffrey L. Schnipper, MD.,MPH., Professor of Medicine, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023P000031; R18HS029366 (AHRQ); 355948 (Other: UCSF IRB)
Record Dates: First submitted 2023-02-07; First posted 2023-02-28 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Diagnostic Errors

STUDY DESIGN:
Intervention Model Description: Interrupted time series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention (usual care) (No Intervention): Patients admitted to study hospitals in the 12 months prior to the start of the intervention
- Intervention (Experimental): Patients admitted to study hospitals during the 36 months of the intervention
  Interventions: Behavioral: ADEPT Program

INTERVENTIONS:
Behavioral: ADEPT Program — Integration of surveillance for diagnostic errors into usual care, benchmarking and sharing of results across hospitals, expert mentoring of quality and safety personnel in change management, pilot testing and refinement of Safety I and Safety II interventions to reduce systemic causes of diagnostic errors and to increase resilience, thus promoting diagnostic excellence.
  Arms: Intervention

SUMMARY:
This study seeks to link a group of hospitals to measure and share the rates of diagnostic errors, to understand underlying causes of diagnostic errors, and develop ways that hospitals, clinicians, and patients can work together to avoid diagnostic errors and harms due to those errors. The investigators will test how data sharing and collaboration improve diagnostic processes and develop approaches which can be sustained into the future. The approach represents a novel application of rigorous outcome adjudication to the problem of inpatient diagnostic errors using a learning health system model.

DETAILED DESCRIPTION:
Many factors contribute to diagnostic errors, but key among them are foundational issues in healthcare: complex and fragmented care systems, the limited time available to providers trying to ascertain a firm diagnosis, and the work systems and cultures that support or impede improvements in diagnostic performance. While approaches to identifying diagnostic errors exist, few studies have linked identification of underlying systemic and structural causes of errors to existing quality improvement programs in hospitals. Even fewer have applied resilience theories or positive deviance approaches to characterize the features of cases where the diagnostic process is optimal and then use those findings to frame health system improvement.

This application builds directly on the investigators' currently funded study - Utility of Predictive Systems in Diagnostic Errors (UPSIDE) - which is defining risk factors, underlying causes, and prevalence of diagnostic errors among patients admitted to hospitals participating in a 55-hospital research collaborative, the Hospital Medicine Reengineering Network (HOMERuN). UPSIDE has developed reference standard approaches to adjudication of diagnostic errors, defined factors associated with errors, and created collaborations with participating sites and national organizations, providing a uniquely powerful opportunity to transform how diagnostic process evaluation programs can be used to improve patient safety.

The overall goal of this Center is to turn the investigators' highly successful multicenter network into a diagnostic error learning health system that will integrate diagnostic error assessments into existing quality and safety programs, provide support and expertise needed to reduce diagnostic errors, and catalyze scientific, personnel, and infrastructure changes which will last beyond the duration of this grant.

To achieve the study's overall goals, the investigators will: 1) Implement a case review infrastructure which can accurately identify diagnostic errors and characterize diagnostic processes among patients suffering inpatient deaths, ICU transfers, or rapid-response team calls taking place at hospitals associated the Hospital Medicine Reengineering Network; 2) Develop site-level audit and feedback and group-wide benchmarking reports of error rates, diagnostic process faults, diagnostic process resilience features and use these data to frame collaboration between existing safety and quality programs at participating sites; 3) Use the data and collaborative model to develop and pilot test interventions based on highest priority findings; and 4) Develop understanding of the program's reach, adoption, implementation, and maintenance, as well feasibility and initial experience with pilot interventions. This project will establish a learning health system which can achieve excellence in diagnosis as an ongoing part of care, a system which can be a model for others as well.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to general medicine services at one of the participating hospitals and who either died during the hospitalization, were transferred to the ICU >= 48 hours after admission, or had a rapid response.

Exclusion Criteria:

* Admitted for a non-medical reason
* Patients coded in the field who are moribund on arrival to the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7200 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Errors | Through hospital discharge, an average of 10 days
  Proportion of patients in each trigger category (death, ICU transfer, rapid response) with an adjudicated diagnostic error.

SECONDARY OUTCOMES:
Harmful Diagnostic Errors | Through hospital discharge, an average of 10 days
  Proportion of patients in each trigger category with diagnostic errors contributing to death, permanent harm, or requiring life-sustaining treatment using NCC-MERP criteria.
Diagnostic process faults | Through hospital discharge, an average of 10 days
  Number of diagnostic process faults per patient, as determined by the DEER taxonomy during adjudication

OTHER OUTCOMES:
Reach | Duration of the program (3 years)
  Description of hospitals, teams, or units where our diagnostic error measurement methodology is built into usual care (Aim 1), where benchmarking data are incorporated into usual care (Aim 2), and whether and which pilot interventions are adopted (Aim 3) compared with those where they are not adopted, and a description of patients who receive patient-level interventions (Aim 3) compared with those who do not.
Adoption | Duration of the program (3 years)
  Number and types of audit/feedback, benchmarking, and Safety I and Safety II interventions adopted at each site, as well as units, teams, and clinician types that do and do not adopt interventions.
Implementation | Duration of the program (3 years)
  Proportion of patients in each trigger population who undergo adjudication for diagnostic error, the number of surveys administered and interviews conducted with medical teams (in the presence of error and for good catches), the number of benchmarking reports produced, the number of audit/feedback sessions conducted, and (if they can be tracked) the proportion of patients who receive patient-level interventions.
Maintenance | Duration of the program (3 years) plus 6 months
  Proportion of patients in each trigger category (death, ICU transfer, rapid response) with an adjudicated diagnostic error 6 months after after the end of collaborative calls with sites.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Auerbach, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - Brigham & Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided